CLINICAL TRIAL: NCT05964972
Title: Impact of an Automatic Alert Device on the Occurrence of Nocturnal Falls in Nursing Home Residents
Acronym: NOCTUSAFE
Status: Terminated | Type: Observational
Why Stopped: lack of patients
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 19-145
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Fall Patients

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Impact of an automatic alert device on the occurrence of nocturnal falls in nursing home residents Measurement of the number of nocturnal falls between 8 p.m. and 8 a.m. per registered resident in the 6 months preceding use of the device compared with the number of nocturnal falls in the 6 months after installation of the device.

ELIGIBILITY:
Inclusion Criteria:

* Resident of the elderly nursing home (EHPAD LES ORCHIDEES).
* Repeated nocturnal falls (more than 2 falls at night between 8 p.m. and 8 a.m.) during the last 12 months.
* Consent of the resident or his legal representative.
* Signature of informed consent
* French-speaking resident.

Exclusion Criteria:

* Refusal to participate in the study.
* Resident exclusive day faller.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fallers
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
number of falls | 6 month preceding and 6 month after
  Measurement of the number of nocturnal falls between 8 p.m. and 8 a.m. per registered resident in the 6 months preceding use of the device compared with the number of nocturnal falls in the 6 months after installation of the device.

CONTACTS AND LOCATIONS:
Locations (1):
- Ehpad Les Orchidees, Cagny, France

IPD SHARING:
Plan to Share IPD: No